CLINICAL TRIAL: NCT06808919
Title: The Effect of Different Exercise Approaches on Passive Mechanical Properties of Hamstring and Quadriceps Muscles, Strength and Jumping Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Selim Mahmut GÜNAY, Doctor of Physical Therapy, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019-19/21
Record Dates: First submitted 2025-01-26; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Healty; Sedantary Activity; Young; Female
Keywords: Stiffness; thickness; elastography; vibration; exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Whole Body Vibration Exercise (Experimental): Whole body vibration exercises were conducted utilizing a specialized exercise platform. The participants underwent a prescribed exercise protocol involving both static and dynamic exercises on the designated platform. Specifically, static squats at a 30º angle, dynamic deep squats ranging from 30 to 60º, toe raises, weight transfer maneuvers during squats, as well as static and dynamic squat exercises performed unilaterally were implemented as part of the program. Each exercise was performed for 30-50 s with a frequency ranging from 30-45 Hz and an amplitude of 2 mm. The exercise regimen was structured to comprise three sets, with a designated three-minute inter-set rest interval. Physical exercise sessions were conducted on a weekly basis, with a duration ranging from 30 to 45 minutes. The intensity and duration of the exercises were progressively adjusted based on the adherence.
  Interventions: Other: Whole Body Vibration Exercise
- Aerobic Exercise (Experimental): Aerobic exercise group were directed to engage in running activity on a conventional treadmill. The participants engaged in aerobic exercise, specifically moderate-to-high-intensity running at 65-80% of their maximal heart rate, for durations of 30-45 minutes per session, three times weekly. Heart rate was monitored with a portable pulse oximetry device.
  Interventions: Other: Aerobic Exercise
- Strengthening Exercise (Experimental): Strengthening exercise group, participants engaged in various lower extremity strengthening activities such as straight leg raises, abduction and adduction movements, knee flexion-extension, ankle plantar-dorsiflexion exercises. These exercises were performed both on a bed and in standing positions, utilizing resistance exercise bands.
  Interventions: Other: Strengthening Exercise
- Control Group (No Intervention): The participants continued their daily lives without any exercise practice until the end of the study.

INTERVENTIONS:
Other: Whole Body Vibration Exercise — The participants underwent a prescribed exercise protocol involving both static and dynamic exercises on the designated platform. Specifically, static squats at a 30º angle, dynamic deep squats ranging from 30 to 60º, toe raises, weight transfer maneuvers during squats, as well as static and dynamic squat exercises performed unilaterally were implemented as part of the program
  Other Names: WHole Body Vibration
  Arms: Whole Body Vibration Exercise
Other: Aerobic Exercise — The participants assigned to the aerobic exercise group were directed to engage in running activity on a conventional treadmill. The participants engaged in aerobic exercise, specifically moderate-to-high-intensity running at 65-80% of their maximal heart rate, for durations of 30-45 minutes per session, three times weekly. Heart rate was monitored with a portable pulse oximetry device.
  Arms: Aerobic Exercise
Other: Strengthening Exercise — Strengthening group, participants engaged in various lower extremity strengthening activities such as straight leg raises, abduction and adduction movements, knee flexion-extension, ankle plantar-dorsiflexion exercises. These exercises were performed both on a bed and in standing positions, utilizing resistance exercise bands.
  Arms: Strengthening Exercise

SUMMARY:
The mechanical characteristics play a crucial role in sustaining daily life activities and facilitating participation in sport activities and exercises demanding a diverse range of motion. Furthermore, it is postulated that the mechanical composition of the muscle could impact the minimal energy expenditure, perceived exertion, and risk of injury during physical activities. This study aims to examine the effects of various exercise approaches, including aerobic exercise, strength training, and whole-body vibration, on the passive mechanical properties of muscle tissue.

DETAILED DESCRIPTION:
Exercise applications are utilized in the maintenance of functional status, enhancement of performance, and prevention of injuries in healthy individuals while also serving therapeutic purposes in pathological conditions. Exercise programs implemented in both healthy individuals and those with disabilities have the potential to offer clinical and functional benefits, leading to physiological changes and mechanical adaptations within the muscle.The enhancement of muscle strength, endurance, and functional performance is observed in accordance with the individuals' physical fitness level and the type of exercise program undertaken. One additional determinant influencing performance is the passive mechanical properties of the muscle. The phrase "passive mechanical properties" denotes the mechanical properties exhibited by skeletal muscles in a state of quiescence, i.e., devoid of voluntary contraction. The passive mechanical properties of muscle encompass properties such as muscle tone, stiffness, thickness, and elasticity. Furthermore, it is postulated that the mechanical composition of the muscle could impact the minimal energy expenditure, perceived exertion, and risk of injury during physical activities. When implemented in either isolated or combined programs, exercises focusing on strengthening, stretching, and aerobic activities can have an impact on muscle mechanics.8,9 Within scholarly literature, there exist investigations that suggest a limited impact on the mechanical properties of muscles following exercise, alongside findings that demonstrate consistent exercise does not induce alterations in muscle stiffness.

Within academic discourse, it is established that power, force, and movement speed represent pivotal elements in elucidating superior performance at an advanced level. Physical fitness parameters, as demonstrated determinants of performance, exhibit direct correlation with muscle structure. The aim of this study was to examine the impact of various exercise approaches, including aerobic, strength training, and whole-body vibration, on passive mechanical properties of muscle tissue. Additionally, the study sought to assess how potential alterations in muscle mechanics might manifest in terms of performance outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy and able to engage in the exercise program without any impediments.
* Voluntary participation

Exclusion Criteria:

* Prior surgical interventions.
* Neuromuscular or neurodegenerative disorders.
* Heart failure.
* Cardiac stents.
* Pregnancy.
* Participants who do not meet the above criteria, even if their current health status permits participation in exercise activities.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | Baseline and at Week 4
  Isokinetic testing and rehabilitation systems were utilized to assess muscle strength. An assessment was conducted on the concentric and eccentric forces exerted on the quadriceps femoris and hamstring muscles in the dominant lower extremity. The assessment of concentric strength was conducted within the knee flexion range of 0-90 degrees, while the evaluation of eccentric strength was undertaken in the knee flexion range of 10-90 degrees at a velocity of 60º/sec. The peak torque values acquired from the experiment were utilized as the basis for the analysis.
Horizontal Jump | Baseline and at Week 4
  Test was conducted unilaterally on the dominant lower extremity. Horizontal jump was repeated three times and the average of the measurement results was recorded.
Muscle Stiffness | Baseline and at Week 4
  Changes in muscle stiffness were evaluated through shear wave elastography. The alterations in the stiffness properties of the muscle were documented utilizing an ultrasound device. Measurements were conducted on the dominant lower extremity to evaluate alterations in the muscle stiffness of the quadriceps muscles (vastus medialis obliquus, rectus femoris) and hamstring muscles (biceps femoris, semimembranosus).
Muscle Thickness | Baseline and at Week 4
  Changes in muscle thickness were evaluated through shear wave elastography. The alterations in the thickness properties of the muscle were documented utilizing an ultrasound device. Measurements were conducted on the dominant lower extremity to evaluate alterations in the muscle thickness of the quadriceps muscles (vastus medialis obliquus, rectus femoris) and hamstring muscles (biceps femoris, semimembranosus).

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Uysal O, Delioglu K, Firat T. The effects of hamstring training methods on muscle viscoelastic properties in healthy young individuals. Scand J Med Sci Sports. 2021 Feb;31(2):371-379. doi: 10.1111/sms.13856. Epub 2020 Nov 3. PMID 33084051
- [Background] Blazevich AJ. Adaptations in the passive mechanical properties of skeletal muscle to altered patterns of use. J Appl Physiol (1985). 2019 May 1;126(5):1483-1491. doi: 10.1152/japplphysiol.00700.2018. Epub 2018 Nov 9. PMID 30412028